CLINICAL TRIAL: NCT05983432
Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Efficacy of BL-B01D1 in Subjects With Metastatic or Unresectable Non-Small Cell Lung Cancer and Other Solid Tumors
Brief Title: Evaluate BL-B01D1 in Patients With Metastatic or Unresectable Non-Small Cell Lung Cancer (NSCLC) and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-LUNG-101
Record Dates: First submitted 2023-07-12; First posted 2023-08-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer; Breast Cancer; Esophageal Cancer; Small Cell Lung Cancer; Nasopharyngeal Cancer; Head and Neck Squamous Cell Carcinoma; Prostate Adenocarcinoma; Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Breast Neoplasms; Esophageal Neoplasms; Small Cell Lung Carcinoma; Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 administered Day 1 and Day 8 per cycle (Experimental): BL-B01D1 will be administered on Day 1 and Day 8 by intravenous infusion every 3 weeks
  Interventions: Drug: BL-B01D1
- BL-B01D1 administered Day 1 per cycle (Experimental): BL-B01D1 will be administered on Day 1 via by intravenous infusion every 3 weeks
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — BL-B01D1 will be administered either on a Day 1 or Day 1 Day 8 dosing regimen

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and efficacy of BL-B01D1 in patients with Metastatic or Unresectable Non-Small Cell Lung Cancer (NSCLC) and Other Solid Tumors.

DETAILED DESCRIPTION:
BL-B01D1-LUNG-101 is a global, multi-center, Phase 1 study to evaluate the safety, tolerability, pharmacokinetics , and initial efficacy of BL-B01D1 in participants with metastatic or unresectable NSCLC and Other Solid Tumors.

This study will be conducted in two different dosing schedules (Cohort A and Cohort B) and three parts (dose escalation, dose finding and dose expansion). Cohort A will be dosed on Day 1 and Day 8 of a continuous 21-day treatment cycle. Cohort B will be dosed on Day 1 of a continuous 21-day treatment cycle. Each Cohort has different dose groups.

ELIGIBILITY:
Inclusion criteria:

1. Signed the informed consent voluntarily and agreed to follow the program requirements
2. Either sex
3. Age: ≥18 years
4. Has a life expectancy of ≥3 months
5. Has histologically documented, incurable, locally advanced or metastatic epithelial origin malignant cancer, priority to include the following tumor types: NSCLC, HER2 - breast cancer, esophageal cancer, SCLC, NPC, and HNSCC.

   Has documented locally advanced or metastatic HER2 negative (by immunohistochemistry [IHC], score of 0 or 1) Hormone Receptor (HR) positive (HER2-, HR+) OR HER2 negative (IHC score of 0 to 2) HR negative breast cancer (HER2-, HR-) as per ASCO CAP criteria (ASCO CAP 2023; Wolff et al. 2023), not amenable to curative surgery or radiation with documentation of radiological disease progression while on/after receiving most recent treatment regimen for locally advanced or metastatic disease, must have received 1 prior line of chemotherapy for advanced disease and, when applicable and if approved in that region, a PD-1/PD-L1 inhibitor, either given concurrently or sequentially. When appropriate, must have progression on at least 1 prior line of hormonal therapy with or without a targeted therapy (such as CDK4/6, mTOR, or PI3-K inhibitors) administered for treatment of metastatic disease.

   In Dose Escalation and Dose finding portions of the study, for triple-negative breast cancer (TNBC, HER2-/HR-) participants must have received PARP inhibitors if a BRCA mutation is present and sacituzumab govitecan as second line treatment. Participants who are HER2 low must have received trastuzumab deruxtecan.
6. Agree to provide archived tumor samples (tissue block or slides) from primary or metastatic sites within 2 years. In the event that no archival tissue is available a fresh tissue biopsy is highly encouraged but not mandatory.
7. Has at least one measurable lesion based on RECIST V1.1 (with the exception of Prostate adenocarcinoma cohort, where subjects with bone metastasis are allowed)
8. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 1
9. Toxicity of previous antitumor therapy has returned to level ≤1 as defined by NCI-CTCAE V5.0 (except for asymptomatic laboratory abnormalities such as elevated ALP, hyperuricemia, elevated serum or plasma amylase/lipase, and elevated blood glucose; except for toxicity that the investigator determined to have no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement therapy, etc.)
10. Has no serious cardiac dysfunction, left ventricular ejection fraction ≥50%
11. Has adequate organ function before registration, defined as: a) Marrow Function: Absolute neutrophil count (ANC) ≥1.2×109 /L, Platelet count ≥100×109 /L, Hemoglobin (Hb) ≥90 g/L b) Hepatic function: Total bilirubin（TBIL≤1.5 ULN, AST and ALT without liver metastasis ≤2.5 ULN, AST and ALT with liver metastasis ≤5.0 ULN c) Renal function: Creatinine clearance ≥50 mL/min (According to the Cockcroft and Gault equation)
12. Coagulation function: international normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (APTT) ≤1.5 ULN
13. Urinary protein ≤2+ or ≤1000mg/24 hours
14. Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception during the course of the study and for 7 months for females and 4 months for males after the last dose of study treatment. An additional contraceptive method, such as a barrier method like a condom is required.
15. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and must be nonlactating. Female subjects are considered WOCBP unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman >45 years old in the absence of other biological or physiological causes. In addition, females <55 years old must have a serum follicle stimulating hormone (fsh) level > 40 mIU/mL to confirm menopause.
16. For subjects with NSCLC (EGFR mutation):

    a) Evidence of documented EGFR TKI-sensitizing deletion mutation in EGFR Exon 19 (ex19del) or leucin-arginine substitution point mutation in EGFR Exon 21 (ex21L858R), the serine-isoleucine mutation in EGFR Exon 20 (ex20S768I), the leucine-glutamine substitution mutation in Exon 21 (ex21L861Q), or the glycine substitution (with alanine, cysteine, or serine) mutation in Exon 18 (ex18G719X) at or after the time of disease diagnosis and prior to initiation of treatment.
17. For Triple-Negative Breast Cancer (TNBC, HER2-/HR-):

    a) Histologically or cytologically confirmed and documented locally advanced, recurrent inoperable or metastatic TNBC
18. For Esophageal adenocarcinoma

    a) Has locally advanced or metastatic adenocarcinoma cell carcinoma of the esophagus or esophagogastric junction cancers, not amenable to curative surgery or radiation with documentation of radiological disease progression after one line of fluoropyrimidine and/or platinum-based chemotherapy treatment regimen for locally advanced or metastatic disease.

    NOTE: Prior therapies such as trastuzumab, zolbetuximab, or IOs are allowed in the study.
19. For Prostate adenocarcinoma

    a) Subject has metastatic castration-resistant prostate cancer (mCRPC) after progression on/after an androgen receptor pathway inhibitors (ARPI) treatment, such as abiraterone, enzalutamide, apalutamide and darolutamide.

    Note: No prior chemotherapy including docetaxel is allowed Prior treatment with lutetium Lu 177 vipivotide tetraxetan (Pluvicto) is allowed. Enrollment will be capped for lutetium Lu 177 vipivotide tetraxetan-naive participants at approximately 20 or participants with prior lutetium Lu 177 vipivotide tetraxetan treatment at approximately 20.
20. For NSCLC (EGFR wild type) with squamous histology

    1. Has documented locally advanced or metastatic NSCLC, not amenable to curative surgery or radiation with documentation of radiological disease progression while on/after receiving most recent treatment regimen for locally advanced or metastatic disease with predominantly squamous cell histology
    2. Must have documented negative test results for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK). Must have no known genomic alterations in ROS proto-oncogene 1 (ROS1).
    3. Progressed or intolerant to one line of platinum-based chemotherapy with α-PD-1/L1 monoclonal antibody given either concurrently or sequentially.
21. For NSCLC (EGFR wild type) with adenocarcinoma histology

    1. Has documented locally advanced or metastatic NSCLC, not amenable to curative surgery or radiation with documentation of radiological disease progression while on/after receiving most recent treatment regimen for locally advanced or metastatic disease with predominantly adenocarcinoma histology
    2. Must have documented negative test results for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK). Must have no known genomic alterations in ROS proto-oncogene 1 (ROS1).

    Progressed or intolerant to one line of platinum-based chemotherapy with α-PD-1/L1 monoclonal antibody given either concurrently or sequentially.
22. Ovarian adenocarcinoma

    a) Has histologic documentation of epithelial ovarian, primary peritoneal, or fallopian tube cancer that has progressed or relapsed on or after a previous platinum-containing chemotherapy with or without a PARP inhibitor.

    Note: participants with platinum-sensitive or platinum resistant recurrent ovarian cancer (PSR) are eligible. However, enrollment will be capped for platinum-sensitive or platinum resistant participants at approximately 20 each.

    Prior bevacizumab treatment is allowed.
23. Endometrial carcinoma

    a) Has relapsed, advanced and/or metastatic endometrial carcinoma, who have progressed on or after prior platinum-based chemotherapy with or without immuno-oncology (IO) treatment
24. For Cervical carcinoma Has relapsed, advanced and/or metastatic cervical carcinoma, who have progressed on or after prior platinum-based chemotherapy with or without immuno-oncology (IO) treatment

Exclusion criteria:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other anti-tumor therapy within 2 weeks or 5 half-lives (whichever is shorter) prior to the first administration; major surgery within 4 weeks prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration
2. Participants with history of severe heart disease, such as symptomatic congestive heart failure (CHF) ≥ Grade 2 (CTCAE 5.0), New York Heart Association (NYHA) ≥ Grade 2 heart failure, history of transmural myocardial infarction, unstable angina pectoris etc;
3. Subjects with prolonged QT interval (QTc >470 msec), complete left bundle branch block, Grade 3 atrioventricular block
4. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for Type I diabetes, hypothyroidism that can be controlled only by standard of care treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis)
5. Other malignant tumors were diagnosed within 5 years prior to the first administration with the following exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after radical resection
6. Participants with poorly controlled hypertension by two kinds of antihypertensive drugs (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg)
7. Participants have Grade 3 lung disease defined according to NCI-CTCAE v5.0, a history of interstitial lung disease (ILD)/ pneumonitis
8. Unstable thrombotic events such as deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring therapeutic intervention within the previous 6 months before screening; Infusion set-related thrombosis is excluded
9. Participants with primary tumors in the central nervous system (CNS) and active or untreated CNS metastases and/or carcinomatous meningitis should be excluded. Participants with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and no requirements for corticosteroids 14 days prior to dosing with the investigational product (IP). Participants on low dose corticosteroids (<20 mg prednisone or equivalent/day) may participate.
10. Participants who have a history of allergies to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL-B01D1
11. Participants have a history of autologous or allogeneic stem cell transplantation (Allo-HSCT)
12. Has received treatment with anthracyclines with a cumulative dose exceeding 360 mg/m2
13. Participants with ≥ Grade 2 hypokalemia (low concentration of potassium in the blood) according to CTCAE v5.0 (Grade 1: participant asymptomatic with potassium levels <LLN - 3.0 mmol/L or equivalent)
14. Known Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active Hepatitis B virus infection (HBV-DNA copy number> the lower limit of detection) or active Hepatitis C virus infection (HCV antibody positive and HCV-RNA > the lower limit of detection)
15. Participants with active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis.
16. Received an investigational drug within 4 weeks, or two half-lives (whichever is longer) prior to first dose of study treatment
17. Participants who are pregnant or breastfeeding
18. Other conditions that the investigator believes may make the subject not suitable for participating in this clinical trial.
19. Participants who have received prior therapy with any ADC targeting EGFR and/or HER3 or containing a topoisomerase 1 inhibitor payload (all dose expansion cohorts with exception of TNBC noted below).

    Note: For TNBC dose expansion cohort, participants with prior ADC therapy targeting HER3 and EGFR or a topoisomerase I inhibitor, such as sacituzumab govitecan may be enrolled with Sponsor consultation prior to enrollment
20. For NSCLC EGFRmut:

    1. Participants treated with more than two systemic chemotherapies prior to randomization.

       NOTE: Progression of disease within 12 months after receiving neoadjuvant and adjuvant chemotherapies is considered 1 prior systemic chemotherapy
    2. Previously documented EGFR Exon 20 insertion mutations as primary EGFR mutations
21. For Triple-Negative Breast Cancer (TNBC, HER2-/HR-):

    a) Participants treated with more than two systemic chemotherapies prior to randomization.

    NOTE: Progression of disease within 12 months after receiving neoadjuvant and adjuvant chemotherapies is considered 1 prior systemic chemotherapy
22. For Esophageal Carcinoma a) Participants received more than 1 prior line of systemic chemotherapy therapy for locally advanced or metastatic disease. NOTE: this limit only applies to prior systemic chemotherapy.
23. For Prostate adenocarcinoma:

    a) Prior treatment with systemic chemotherapy.
24. For NSCLC with EGFR WT squamous or adenocarcinoma histology: a) Participants received more than 1 prior line of systemic chemotherapy for locally advanced or metastatic disease
25. For Ovarian Carcinoma a) Participants received more than 1 prior line of systemic chemotherapy. Re-treatment with platinum-based chemotherapy is considered one line of therapy. Prior hormonal therapy is permitted.
26. For Endometrial Carcinoma a) Participants received more than 1 prior line of systemic chemotherapy. Re-treatment with platinum-based chemotherapy is considered one line of therapy. Prior hormonal therapy is permitted.
27. For Cervical Carcinoma a) if received more than 1 prior line of systemic chemotherapy. Re-treatment with platinum-based chemotherapy is considered one line of therapy.

Notes: Re-treatment with platinum-based chemotherapy is considered one line of therapy.

Note: A participant who does not meet this exclusion criterion may be allowed into the study pending the sponsor's approval, based on current accrual within this dose expansion cohort.

Note: There is no limit on the number of prior lines of non-chemotherapy regimens. ADCs with cytotoxic payloads are considered a line of chemotherapy. For any expansion cohorts, if only limited number of patients can be enrolled with 1 prior line of chemotherapy, the Sponsor has the option to allow participants with more than 1 prior line of chemotherapy to be enrolled, upon Sponsor's approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
Participants with Dose-limiting toxicities | One year
  Measuring the number of patients Dose-limiting toxicities (DLTs). A DLT is defined as any of the following events that are not clearly due to the underlying disease or extraneous causes:
  Hematological toxicities:
  * Grade 4 neutrophil count decreased lasting >7 days
  * Grade ≥3 febrile neutropenia
  * Grade ≥3 platelet count decreased with clinically significant hemorrhage.
  Non-Hematological toxicities:
  * Death
  * Hy's law cases
  * Grade ≥3 non-hematological toxicities,
Participants with Serious Adverse Events (SAEs) and treatment-emergent adverse events (TEAEs), | One year
  Measuring the number of patients with serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs)
Participants with abnormal physical examination findings | One year
  Measure the number of participants with abnormal physical examination findings.
Participants with ability to care for themselves, daily activity, and physical activity | One year
  Measure the change in participants with Eastern Clinical Oncology Group (ECOG) Scale of Performance Status. The scale is 0-4 with 0 being the fully active (best outcome) and 4 being completely disabled (worst outcome)
Participants with abnormal ECG reading | One year
  Measure the number of participants with abnormal ECG parameters
Participants with abnormal lab results | One year
  Measure the number of participants with abnormal clinical laboratory values
To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and two or more recommended doses and schedules for recommended dose expansion (RDEs) of BL-B01D1 in metastatic NSCLC | One year
  Determine the highest BL-B01D1 dose level at which ≤33% subjects experience a DLT during the DLT evaluation period and highest BL-B01D1 dose administered in the event and MTD cannot be defined.

SECONDARY OUTCOMES:
Cmax of BL-B01D1 | One year
  Calculate maximum (peak) observed concentration of BL-B01D1
Cmax of anti-EGFR×HER3 antibody | One year
  Calculate maximum (peak) observed concentration of anti-EGFR×HER3 antibody
Cmax of free payload ED-04 | One year
  Calculate maximum (peak) observed concentration of free payload ED-04
Tmax of BL-B01D1 | One year
  Calculate time of maximum observed concentration of BL-B01D1
Tmax of anti-EGFR×HER3 antibody | One year
  Calculate time of maximum observed concentration of anti-EGFR×HER3 antibody
Tmax of free payload ED-04 | One year
  Calculate time of maximum observed concentration of free payload ED-04
AUC(0-8) of BL-B01D1 | One year
  Calculate area under the serum concentration-time curve of BL-B01D1 from time 0 to 8 hours
AUC(0-8) of anti-EGFR×HER3 antibodies | One year
  Calculate area under the serum concentration-time curve of anti-EGFR×HER3 antibodies from time 0 to 8 hours
AUC(0-8) of free payload ED-04 | One year
  Calculate area under the serum concentration-time curve of free payload ED-04 from time 0 to 8 hours
AUC(last) of BL-B01D1 | One year
  Calculate area under the serum concentration-time curve up of BL-B01D1 to the last quantifiable time
AUC(last) anti-EGFR×HER3 antibodies | One year
  Calculate area under the serum concentration-time curve up of anti-EGFR×HER3 antibodies to the last quantifiable time
AUC(last) of free payload ED-04 | One year
  Calculate area under the serum concentration-time curve up of free payload ED-04 to the last quantifiable time
Overall Response Rate (ORR) | One year
  To assess the clinical efficacy of BL-B01D1 as measured by ORR using RECIST criteria v 1.1
Disease Control Rate (DCR) | One year
  To assess the clinical efficacy of BL-B01D1 as measured by DCR using RECIST criteria v 1.1
Time To Response (TTR) | One year
  To assess the clinical efficacy of BL-B01D1 as measured by TTR using RECIST criteria v 1.1
Progression-Free Survival (PFS), | One year
  To assess the clinical efficacy of BL-B01D1 as measured by PFS using RECIST criteria v 1.1
Overall Survival (OS). | One year
  To assess the clinical efficacy of BL-B01D1 as measured by OS using RECIST criteria v 1.1
Antitumor Activity | One year
  To investigate the antitumor activity of BL-B01D1 as evaluated using RECIST Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Zhao, MD, PhD, Study Director — SystImmune Inc.
Locations (39):
- United States (24):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - City of Hope Cancer Center, Duarte, California
  - Chao Family Comprehensive Cancer Care and Ambulatory Care, Irvine, California
  - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - University of California Irvine Medical Center, Orange, California
  - UCLA Santa Monica, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Sara Cannon Research Institute Lake Nona, Orlando, Florida
  - Hematology - Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Head Neck Services, New York, New York
  - PRISMA Health/ITOR, Greenville, South Carolina
  - Sarah Cannon - Tennessee Oncology, Nashville, Tennessee
  - Oncology Consultants, P.A., Houston, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington Fred Hutchinson, Seattle, Washington
- France (4):
  - Centre Léon Bérard, Lyon
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Institut de Cancerologie de Ouest (ICO) - Saint-Herblain, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo
  - IRCCS Istituto Clinico Humanitas, Cancer Center, Rozzano
- National Cancer Center Hospital, Chūōku, Japan
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Beata María Ana, Madrid
  - START Madrid / Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - START Madrid / Centro Integral Oncologico Clara Campal, Madrid
  - START Rioja, Piqueras
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No